CLINICAL TRIAL: NCT01879085
Title: Phase 1b/2 Study of Vorinostat in Combination With Gemcitabine and Docetaxel in Advanced Sarcoma
Brief Title: Study of Vorinostat in Combination With Gemcitabine and Docetaxel in Advanced Sarcoma
Acronym: GemTax
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Melissa Burgess, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Melissa Burgess, MD, Assistant Professor of Medicine Division of Hematology/Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCI# 12-104
Record Dates: First submitted 2013-05-20; First posted 2013-06-17 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Sarcoma
Keywords: advanced; metastatic; unresectable; soft; tissue; sarcomas
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Docetaxel; Gemcitabine; Vorinostat; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination therapy (Experimental): Dose Level\Docetaxel IV\ Gemcitabine IV\Vorinostat PO\Pegfilgrastim 1\75 mg/m2\900 mg/m2\300 mg once daily\6 mg on day 9 2\75 mg/m2\900 mg/m2\200 mg twice daily\6 mg on day 9 3\75 mg/m2\900 mg/m2\300 mg twice daily\6 mg on day 9 4\75 mg/m2\900 mg/m2\400 mg twice daily\6 mg on day 9
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Vorinostat; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 IV given over 60 minutes on day 8 every 21 days (1 cycle)
  Other Names: Taxotere
Drug: Gemcitabine — given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle). For dose level -2, given over 67.5 minutes at 10 mg/m2/min
  Other Names: Gemzar
Drug: Vorinostat — given orally at the specified dose levels (either 300 mg/daily or 200 mg twice per day) on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle)
  Other Names: Zolinza
Drug: Pegfilgrastim — administered on day 9 subcutaneously at 6 mg
  Other Names: Neulasta

SUMMARY:
This is a Phase Ib/II experimental, open-label, dose escalation, active treatment study designed to determine the safety, tolerability, and recommended dose of the combination.

During the Phase 2 portion of the study, we will assess progression-free survival (PFS), overall survival (OS),overall response rate (ORR), correlative endpoints, DNA methylation measured by microarray, and expression level of the genes as measured by microarray

DETAILED DESCRIPTION:
Phase 1b

* To determine the dose of vorinostat that can be safely combined with gemcitabine and docetaxel in patients with advanced sarcomas.
* To characterize the Pharmacokinetics (PK) and Pharmacodynamics (PD) of vorinostat when combined with gemcitabine and docetaxel in patients with advanced sarcomas (Exploratory Aim).

Phase 2

* To determine the safety and efficacy of gemcitabine and docetaxel in combination with vorinostat in patients with advanced sarcomas. The hypothesis is that gemcitabine and docetaxel + vorinostat will be safe and will improve the 6-months progression-free rates (PFR) of the combination by 20% (from 20% to 40%).
* To determine the objective response rate, progression-free, and overall survival of patients with advanced sarcomas treated with gemcitabine and docetaxel + vorinostat;
* To develop a predictive molecular signature of response to treatment in advanced sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed soft tissue sarcoma with evidence of metastatic or unresectable disease.
* Patients must have measurable disease by RECIST 1.1.
* Up to 32 prior cytotoxic chemotherapy regimens in the metastatic setting are allowed. Adjuvant chemotherapy or targeted therapy will not be considered a prior line of treatment.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/µL
  * absolute neutrophil count ≥1,500/µL
  * platelets ≥100,000/µL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤1.5 X institutional upper limit of normal (ULN)
  * creatinine ≤1.5 X institutional upper limit of normal (ULN)
* Peripheral neuropathy, if present, should be ≤grade 1.
* Women of Child bearing potential MUST use contraceptives.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* The following specific histologic subtypes of soft tissue sarcomas will be excluded: GIST, Kaposi's sarcoma, mesothelioma, dermatofibrosarcoma, chordoma, alveolar soft-part sarcoma. Also, all bone sarcomas are excluded including Ewing's sarcoma, osteosarcoma, GIST, low grade chondrosarcoma, and chordoma.
* Patients who have had treatment with chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting study treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, docetaxel, vorinostat, or G-CSF.
* Patients who have received and progressed on the combination of gemcitabine and docetaxel in the metastatic setting.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and breastfeeding women
* Patients taking concomitant HDAC inhibitors.
* HIV-positive patients on combination antiretroviral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Burgess, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analysis of Phase 2 group includes (6) patients who enrolled to the Phase 1b group at Dose Level 1.
Groups:
- Dose Level 1; Phase 2: Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle). For dose level -2, Gem will be given over 67.5 minutes at 10 mg/m2/min.
  Vorinostat: given orally at Dose level 1 (300 mg/day) on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
- Dose Level 2: Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle). For dose level -2, Gem will be given over 67.5 minutes at 10 mg/m2/min.
  Vorinostat: given orally at Dose level 2 (200 mg twice/day) on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
Period: Phase 1b
Arm/Group | Dose Level 1 | Dose Level 2 | Phase 2
Started | 6 | 6 | 0
Completed | 6 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Dose Level 1 | Dose Level 2 | Phase 2
Started | 6 | 0 | 25
Completed | 6 | 0 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Dose Level 1:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: 300 mg daily given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
- Dose Level 2: Dose Level 2:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: 200 mg twice daily given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 31 | 6 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.68 (15.16) | 50.50 (17.03) | 55.03 (15.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 3 | 24
  Male | 10 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 30 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 27 | 6 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose of Vorinostat
Description: Recommended Phase ll dose of vorinostat that can be safely combined with gemcitabine and docetaxel. Gemcitabine and docetaxel were given at a fixed dose while vorinostat was dose-escalated using a standard '3+3' design. Dose-limiting toxicity (DLT) is defined as specific study drug-related events experienced during Cycle 1; only DLTs observed in a patient during the first cycle of treatment will be used for the dose escalation decision.
Time Frame: During Cycle 1 of treatment
Population: Patients treated with combination therapy.
Measure: Number; unit: mg/day of Vorinostat
Groups:
- Combination Therapy: Docetaxel + Gemcitabine + Vorinostat + Pegfilgrastim: Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle). For dose level -2, Gem will be given over 67.5 minutes at 10 mg/m2/min.
  Vorinostat: given orally at either 300 mg/day, on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
Arm/Group | Combination Therapy: Docetaxel + Gemcitabine + Vorinostat + Pegfilgrastim
Number analyzed (Participants) | 12
mg/day of Vorinostat | 300

2. Primary Outcome: Six-month Progression-free Survival (PFS)
Description: Proportion of participants whose disease does not progress within 6 months of start of treatment (number of patients without progressive disease/total number of patients). Per RECIST v1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 6 months (per patient)
Population: Patients that received combination therapy that were evaluable for response to treatment.
  Note: Six of the twelve patients enrolled to the Phase 1b group at Dose Level 1 / RP2D were analyzed with the Phase 2 group due to same dose level of vorinostat.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Phase 2: Dose Level 1:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: RP2D - 300 mg daily given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
Arm/Group | Phase 2
Number analyzed (Participants) | 31
proportion of participants | 0.473 [0.325 to 0.69]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Number of patients with Complete response [CR] + partial response [PR], per RECIST v1.1 criteria . Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. For non-target lesions: Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10mm short axis);PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Up to 7 years and 7 months
Population: Patients that received combination therapy. Note: Six of the twelve patients enrolled to the Phase 1b group at Dose Level 1 / RP2D were analyzed with the Phase 2 group due to same dose level of vorinostat.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Dose Level 1:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: RP2D - 300 mg/day given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
Arm/Group | Phase 2
Number analyzed (Participants) | 31
Participants | 7

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The median length of time from the beginning of study treatment that patients remain alive without progression of their disease (cancer). Per RECIST v1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 7 years and 7 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2
Number analyzed (Participants) | 31
months | 5.552361 [2.694045 to 12.41889]

5. Secondary Outcome: One-year Progression-free Survival (PFS)
Description: Proportion of participants whose disease does not progress within one year of start of treatment (number of patients with progressive disease/total number of patients). Per RECIST v1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. For non-target lesions, PD: Unequivocal progression of existing non-target lesions. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to one year (per patient)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 31
proportion of participants | 0.304 [0.177 to 0.523]

6. Secondary Outcome: Overall Survival (OS)
Description: The median length of time from the start of treatment that diagnosed study participants remain alive.
Time Frame: Up to 7 years and 7 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2
Number analyzed (Participants) | 31
months | 11.92608 [10.05339 to 20.33676]

7. Secondary Outcome: Six-month Overall Survival (OS)
Description: Proportion of participants alive at six months from the start of treatment.
Time Frame: Up to 6 months (per patient)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 31
proportion of participants | 0.742 [0.603 to 0.913]

8. Secondary Outcome: One-year Overall Survival (OS)
Description: Proportion of participants alive at one year from the start of treatment.
Time Frame: Up to one year (per patient)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Phase 2
Number analyzed (Participants) | 31
proportion of participants | 0.477 [0.328 to 0.692]

ADVERSE EVENTS:
Time Frame: Both Adverse Events and All-Cause Mortality were assess continuously over a duration of time up to 7 years and 7 months (for the population).
Description: Additional information: Six of the twelve patients enrolled to the Phase 1b group at Dose Level 1 / RP2D were analyzed with the Phase 2 group due to same dose level of vorinostat.
Groups:
- Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 300 mg/Day: Dose Level 1:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: 300 mg daily given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
- Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 200 mg Twice/Day: Dose Level 2:
  Docetaxel: 75 mg/m2 IV over 60 minutes on day 8 every 21 days (1 cycle).
  Gemcitabine: given on days 1 and 8 at 900 mg/m2 IV over 90 minutes (fixed dose infusion rate at 10 mg/m2/min) every 21 days (1 cycle).
  Vorinostat: 200 mg twice daily given orally on days -1 to +2 and days +7-9 every 21 days (treatment for 3 days starting one day prior to chemotherapy on every cycle).
  Pegfilgrastim: Administered on day 9 subcutaneously at 6 mg.
Arm/Group | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 300 mg/Day | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 200 mg Twice/Day
All-Cause Mortality (participants affected / at risk) | 26/31 | 5/6
Serious Adverse Events (participants affected / at risk) | 19/31 | 3/6
Other Adverse Events (participants affected / at risk) | 31/31 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 300 mg/Day (N=31) | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 200 mg Twice/Day (N=6)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Fever (General disorders) | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Investigations - Other, specify (Investigations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Malaise (General disorders) | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 0
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Uspecified (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 300 mg/Day (N=31) | Docetaxel + Gemcitabine + Pegfilgrastim + Vorinostat 200 mg Twice/Day (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Activated partial thromboplastin time prolonged (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 10 | 3
Alkaline phosphatase increased (Investigations) | 19 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 2
Anemia (Blood and lymphatic system disorders) | 30 | 6
Anorexia (Metabolism and nutrition disorders) | 13 | 1
Anxiety (Psychiatric disorders) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 12 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bloating (Gastrointestinal disorders) | 2 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 10 | 1
Blood bilirubin increased (Investigations) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 6 | 1
Chills (General disorders) | 5 | 0
Cholesterol high (Investigations) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 18 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Creatinine increased (Investigations) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Delirium (Psychiatric disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Depression (Psychiatric disorders) | 8 | 4
Diarrhea (Gastrointestinal disorders) | 16 | 0
Dizziness (Nervous system disorders) | 5 | 0
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0
Dysesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 6 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 1
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 17 | 3
Endocrine disorders - Other, specify (Endocrine disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Eyelid function disorder (Eye disorders) | 1 | 0
Fatigue (General disorders) | 22 | 4
Fever (General disorders) | 6 | 2
Flu like symptoms (General disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 1
Gait disturbance (General disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 9 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 12 | 0
Headache (Nervous system disorders) | 8 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 7 | 1
Hypernatremia (Metabolism and nutrition disorders) | 8 | 2
Hypertension (Vascular disorders) | 16 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 26 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 18 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 1
Hyponatremia (Metabolism and nutrition disorders) | 26 | 6
Hypoparathyroidism (Endocrine disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 5
Hypotension (Vascular disorders) | 4 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Immune system disorders - Other, specify (Immune system disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 2 | 5
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 | 0
INR increased (Investigations) | 5 | 1
Insomnia (Psychiatric disorders) | 8 | 3
Investigations - Other, specify (Investigations) | 30 | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 26 | 5
Lymphocyte count increased (Investigations) | 3 | 0
Malaise (General disorders) | 6 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 10 | 0
Movements involuntary (Nervous system disorders) | 1 | 1
Mucosal infection (Infections and infestations) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 22 | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 6 | 0
Neutrophil count decreased (Investigations) | 17 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pain (General disorders) | 18 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Pancreatic enzymes decreased (Investigations) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Platelet count decreased (Investigations) | 27 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 0
Rash pustular (Infections and infestations) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 14 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 13 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Vascular disorders - Other, specify (Vascular disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Weight gain (Investigations) | 2 | 0
Weight loss (Investigations) | 4 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 20 | 2
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Personality Change (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT01879085/Prot_SAP_000.pdf